CLINICAL TRIAL: NCT07204912
Title: Evaluation of a Neural-Controlled Powered Prosthesis Across Diverse Real-World Tasks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2503001589
Record Dates: First submitted 2025-06-16; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Transfemoral Amputation
Keywords: Transfemoral Amputation; Bionic Prosthesis; Knee Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MIT Powered Leg (Experimental): Subjects wears the MIT powered knee-ankle prosthesis.
  Interventions: Device: MIT Powered Leg
- Prescribed prosthesis (No Intervention): Subjects wears their prescribed prosthesis.

INTERVENTIONS:
Device: MIT Powered Leg — MIT powered knee prosthesis developed by the MIT Biomechatronics Group.
  Arms: MIT Powered Leg

SUMMARY:
The purpose of this study is to evaluate the performance and adaptability of a neural-controlled powered knee or ankle prosthesis across diverse real-world mobility tasks. This research aims to assess how compare the sense of embodiment with the device, symmetry, and stability of a person with an lower-extremity amputation walking with a bionic prosthesis and their prescribed prosthesis. Findings from this study will inform future developments in bionic prosthesis design with optimal integration with the human body, with the goal of improving prosthetic integration into daily life.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 18-70.
* The patient must have a unilateral transfemoral amputation .
* The patient must have the ability to ambulate at variable cadence (an expected lower extremity prosthesis functional level of K3 or above).
* The patient must have adequate socket to support the device.

Exclusion Criteria:

* Women who are pregnant.
* Severe co morbidity, atypical skeletal anatomy, or poor general physical/mental health that, in the opinion of the Investigator, will not allow the subject to be a good study candidate (i.e. other disease processes, mental capacity, substance abuse, shortened life expectancy, vulnerable patient population, BMI >40, etc.).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-31 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Kinematic and Kinetic Measures of Lower-Limb Biomechanics | An average of 2 sessions in the span of 1 week
  Quantitative analysis of lower-limb biomechanics, including joint angles, ground reaction forces, joint torques, and mechanical power during level-ground walking, stair negotiation, and other functional tasks. Outcomes will be assessed using a motion capture system (e.g., Vicon), instrumented force plates, and embedded prosthesis sensors to evaluate gait symmetry, stability, and mechanical efficiency.
Spatiotemporal Gait Parameters | An average of 2 sessions in the span of 1 week
  Evaluation of spatiotemporal gait parameters during ambulation with the powered prosthesis. Specific measures include stride length, cadence, walking speed, and stance-to-swing ratio. Parameters will be obtained using a motion capture system (e.g., Vicon) and an instrumented walkway. Data will be analyzed to assess functional walking ability and compared to normative or baseline values
Assessment of Patient Ability to Control each Joint of the Prosthesis | An average of 2 sessions in the span of 1 week
  Assessment of volitional control of the powered knee and ankle joints via neural signals from the residual limb. Participants will perform isolated joint control trials in seated positions. Outcomes include joint command accuracy, latency, and repeatability, evaluated using surface electromyography (EMG) and motion capture. These measures will quantify the participant's ability to intentionally control each prosthetic joint.

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Herr, Principal Investigator — MIT Media Lab
Locations (1):
- MIT Media Lab, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Subject confidentiality.